CLINICAL TRIAL: NCT07307404
Title: Web-based Platform for Nutrition Management in Patients With Cancer: A Randomized Clinical Trial
Brief Title: Web-based Platform for Nutrition Management in Patients With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xingchen Peng (Other)
Responsible Party: Sponsor-Investigator, Xingchen Peng, PhD, Professor, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-2316
Record Dates: First submitted 2025-11-17; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Nutrition
Keywords: cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Self-Intervention: During the period of staying at home, patients use the app developed by the team for self-intervention, including dietary monitoring and check-ins, nutritional risk assessment, learning of educational knowledge, and online expert consultations.
  Community Intervention: When nutritional risks are detected, pop-up alerts will notify patients to communicate with the community management team. Patients can seek basic nutritional consultations and receive advice from the community management team. If necessary, the management team will refer patients to relevant higher-level hospital outpatient clinics for further care. If patients experience other issues related to their primary condition, the community management team will refer them to community healthcare providers for consultation and treatment.
  The community will also organize thematic lectures on nutritional management for cancer patients, with oncologists and nutritionists providing regular voluntary consultatio
  Interventions: Other: nutrtion care based on app
- standard care (No Intervention): standard nutrtion care

INTERVENTIONS:
Other: nutrtion care based on app — Self-Intervention: During the period of staying at home, patients use the app developed by the team for self-intervention, including dietary monitoring and check-ins, nutritional risk assessment, learning of educational knowledge, and online expert consultations.
  Community Intervention: When nutritional risks are detected, pop-up alerts will notify patients to communicate with the community management team. Patients can seek basic nutritional consultations and receive advice from the community management team. If necessary, the management team will refer patients to relevant higher-level hospital outpatient clinics for further care. If patients experience other issues related to their primary condition, the community management team will refer them to community healthcare providers for consultation and treatment.
  The community will also organize thematic lectures on nutritional management for cancer patients, with oncologists and nutritionists providing regular voluntary consultation
  Arms: intervention group

SUMMARY:
It is crucial to promptly identify nutritional issues in these patients within the community and provide them with dietary guidance, nutritional counseling, and support. This study will be conducted in communities in Chengdu, Sichuan. Community management teams will register oncology patients, collecting information such as demographic data, tumor type, stage, specific treatment plan, treatment hospital, regularity of hospital admissions, and frequency of independent smartphone use. Registered patients will be screened based on inclusion and exclusion criteria. For those who meet the criteria, the community management team will contact them and recommend the use of a dedicated app developed by the research team. An initial nutritional assessment will also be conducted. Patients identified with nutritional risks will be directly referred to the research team's clinical nutritionists for face-to-face consultations. After additional tests, such as body composition analysis, necessary nutritional education and stepwise nutritional interventions will be provided. These patients will also use the app for dietary monitoring and nutritional guidance. For patients without nutritional risks, the app will be recommended for daily questionnaire completion and activity tracking.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed malignant tumor;
* PG-SGA score of 4-9 points;
* Age: ≥18 years, with an expected survival time of more than 1 year;
* Possesses adequate cognitive and reading abilities to complete questionnaires and use the APP.

Exclusion Criteria:

* Presence of neurological or psychiatric disorders affecting cognitive function, including central nervous system metastasis of tumors;
* Suffering from conditions severely impacting digestion, metabolism, or food intake;
* Patients in the cachexia stage or refractory cachexia phase.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
body weight change | baseline, pre-intervention；every 2 weeks after randomization until 6 moths.
  change of body weight during the trail

SECONDARY OUTCOMES:
PG-SGA | baseline, pre-intervention；every 2 weeks after randomization until 6 moths.
  assessed using the PG-SGA score
NRS2002 | baseline, pre-intervention；every 2 weeks after randomization until 6 moths.
  using nutrition risk screening [NRS 2002]

OTHER OUTCOMES:
EORTC QLQ C30 | baseline, pre-intervention；every 4 weeks after randomization until 6 moths.
  using Quality-of-Life Questionnaire Core 30
caregiver burden | baseline, pre-intervention；every 4 weeks after randomization until 6 moths.
  using the 12-Item Zarit Burden Interview [ZBI]
psychology characteristics | baseline, pre-intervention；every 4 weeks after randomization until 6 moths.
  Hospital Anxiety and Depression Scale [HADS]

CONTACTS AND LOCATIONS:
Locations (1):
- West China hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided